CLINICAL TRIAL: NCT02023060
Title: Functional and Quality of Life Improvement Following Transcatheter Heart Valve Implantation
Status: Recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-13-0685-IB-CTIL
Record Dates: First submitted 2013-12-09; First posted 2013-12-30 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-06

CONDITIONS: Trans Catheter Aortic Valve; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective is to observe trends in patient characteristics and outcomes after aortic or mitral transcatheter heart valve replacement over time.

DETAILED DESCRIPTION:
To observe trends in patient characteristics and outcomes after aortic or mitral transcatheter heart valve replacement over time.

ELIGIBILITY:
Inclusion Criteria:

1. Subject selected for transcatheter heart valve replacement
2. Signed informed consent to participate in the study

Exclusion Criteria:

1. Inability to sign written informed consent.
2. Pregnancy or breast feeding (women of childbearing potential will have a serum or urine pregnancy test).

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with severe aortic or mitral valve dysfunction (stenosis or regurgitation) selected for transcatheter aortic or mitral valve replacement
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-11; Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome of patients undergoing transcatheter valve replacement | 12 months
  Mortality, change in New York Heart Association class, change in ejection fraction.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Barbash, MD, Study Chair — Sheba Medical Center, Tel Hashomer
Locations (5):
- Israel (5):
  - Hadassah Medical Center, Jerusalem
  - Shaarei Zedek amedical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Medical Center, Tel Aviv

REFERENCES:
- [Derived] Zusman O, Barbash MI, Guetta V, Finkelstein A, Assali A, Segev A, Orvin K, Barsheshet A, Younis A, Witberg G, Kornowski R, Danenberg H, Landes U. Predicting the risk of late futile outcome after transcatheter aortic valve implantation. Catheter Cardiovasc Interv. 2020 Dec;96(7):E695-E702. doi: 10.1002/ccd.28761. Epub 2020 Feb 5. PMID 32022390
- [Derived] Brodov Y, Konen E, Di Segni M, Samoocha D, Chernomordik F, Barbash I, Regev E, Raanani E, Guetta V, Segev A, Fefer P, Glikson M, Goitein O. Mitral Annulus Calcium Score. Circ Cardiovasc Imaging. 2019 Dec;12(1):e007508. doi: 10.1161/CIRCIMAGING.117.007508. PMID 30636515